CLINICAL TRIAL: NCT01453595
Title: A Phase 1b/2 Study of BEZ235 in Patients With Advanced Renal Cell Carcinoma (RCC)
Brief Title: BEZ235 in Patients With Advanced Renal Cell Carcinoma (RCC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Given the number of toxicities seen and the difficulty with patient retention in the dose escalation portion, the sponsor decided to close the trial.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-080
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Renal Cancer
Keywords: Kidney; renal cell carcinoma; BEZ235; 11-080
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — dactolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BEZ235 (Experimental): This is a single-institution, open label, single-arm Phase 1b/2 trial of BEZ235 in patients with advanced RCC. The study will be conducted in two phases:
  Phase 1b: dose-escalation will be performed to determine the maximally tolerated dose (MTD) of twice daily BEZ235 to use in Phase 2 (RP2 dose).
  Phase 2: subjects with clear cell who have experienced disease progression on prior first or second-line mTOR targeted therapy will be treated on the MTD of twice daily BEZ235.
  Interventions: Drug: BEZ235

INTERVENTIONS:
Drug: BEZ235 — BEZ235 will be taken orally twice daily starting on Day 1, Cycle 1, self-administration will continue twice daily on a continuous schedule with cycle length defined as 28 days. Increasing dosing levels of BEZ235 will be studied sequentially (beginning with Dose Level 1, BEZ235 400mg by mouth twice daily) as per the treatment noted below.
  Cohort-1a BEZ235 300 mg by mouth twice daily Cohort 1 BEZ235 400 mg by mouth twice daily Cohort 2 BEZ235 600 mg by mouth twice daily Cohort 3 BEZ235 800 mg by mouth twice daily

SUMMARY:
This study tests a new medication for treatment of kidney cancer, called BEZ235. This medication works by blocking several mechanisms that the cancer needs to grow and survive. By blocking these mechanisms, the medication can thus suppress further growth of the cancer, possibly kill cancer cells. Older kidney cancer medications (such as temsirolimus [Torisel®] or everolimus [Afinitor®]) typically only block one mechanism in cancer cells, so the investigators think that BEZ235 may work even better against kidney cancer.

The purpose of the first part of this study is to test the safety of giving BEZ235 at different doses. The investigators are trying to find a safe dose of BEZ235 and want to find out what effects, good and/or bad, it has on the patient and the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced renal cell carcinoma. Advanced disease is defined as unresectable, locally recurrent disease or metastatic disease. This must by confirmed by MSKCC pathology review with the following requirements:
* Phase 1b: Any histologic subtype of RCC.
* Phase 2: clear cell type RCC or predominant clear cell component.

Patients will be screened for prior systemic therapies:

* Phase 1b: Any prior therapy.
* Phase 2: Progression of disease on at least one prior treatment with an mTOR inhibitor (such as everolimus, temsirolimus, ridaforolimus). Other prior systemic therapies including VEGF directed therapy (e.g. sunitinib, sorafenib, bevacizumab) and immunotherapy (e.g. IL-2, interferon-α) are also permitted. Evidence of unidimensionally measurable disease per RECIST 1.1 (Eisenhauer, Therasse et al. 2009).
* Resolution of all acute toxic effects of prior systemic treatments, radiotherapy or surgical procedures to NCI CTCAE Version 4.0 grade ≤1.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, which is not declining during the last 2 weeks.
* 18 years of age or older.

Adequate organ function as defined by the following criteria:

* Absolute neutrophil count (ANC) ≥1,000/μL
* Platelets ≥100,000/μL
* Hemoglobin ≥9.0 g/dL
* Serum calcium ≤12.0 mg/dL
* Serum creatinine ≤1.5 x upper limit of normal (ULN); if this is exceeded, estimated creatinine clearance must be ≥ 30 ml/min
* Total serum bilirubin ≤ 1.5 x ULN (in patients with known Gilbert Syndrome, a total bilirubin of ≤ 3 x ULN, with direct bilirubin ≤ 1.5 x ULN)
* Serum aspartate transaminase (AST) and serum alanine transaminase (ALT)

  ≤3 x ULN (≤5 x ULN in the setting of hepatic metastases)
* INR ≤ 2. (Anticoagulation with warfarin is contraindicated)
* Fasting plasma glucose (FPG) ≤ 140mg/dL
* HgbA1c ≤ 8%
* Fasting serum cholesterol ≤300 mg/dL, fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication. Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to undergoing study screening procedures.
* Subject's willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Patients who have received prior treatment with a P13K inhibitor (Phase 2 portion only).
* Patients within 28 days post major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) or significant traumatic injury.
* Patients who had radiation therapy within 28 days prior to start of study treatment (palliative radiotherapy to bone lesions allowed if completed 2 weeks prior to study treatment start).
* Patients who have received chemotherapy, immunotherapy or other investigational agents ≤ 2 weeks prior to study treatment start.

Patients currently receiving medications known to be inducers or moderate / strong inhibitors of CYP3A4 (see table 9.2 for a list) Patients must discontinue such medications ≥ 7 days prior to initiation of study treatment.

* Patients currently receiving medications with a significant risk to induce Torsades de Pointes
* Patients who are currently receiving treatment with warfarin sodium (Coumadin®). If treatment is discontinued or switched to an alternate anticoagulant prior to enrollment, INR within ≤48h prior to study initiation has to return to ≤ 2 x ULN.
* Patients receiving chronic treatment with systemic corticosteroids or other immunosuppressive agents (inhaled or topical steroids are allowed)
* Patients with evidence or history of central nervous system (CNS) metastases or spinal cord compression, unless prior treatment with surgery or radiotherapy AND no progression of CNS disease within 6 months prior to enrollment. Patients must not be receiving chronic corticosteroid therapy for CNS metastases.
* Patients who have a history of severe medical conditions or other conditions that could affect their participation in the study such as:
* symptomatic intrinsic lung disease requiring oxygen supplementation at baseline
* uncontrolled hypertension (i.e., SBP>180 mmHg or DBP >100mmHg)
* any active (acute or chronic) or uncontrolled infection/disorders that impair the ability to evaluate the patient or for the patient to complete the study
* liver disease such as cirrhosis or decompensated liver disease.
* Impairment of gastrointestinal function that may impair absorption of BEZ235 (e.g. ulcerative diseases, uncontrolled nausea/vomiting; diarrhea ≥ grade 2; malabsorption syndromes after prior small-bowel resection)
* Immunocompromised patients and/or history of HIV seropositivity

Patients with prior or current cardiac problems including:

* History of unstable angina pectoris (at any time), symptomatic congestive heart failure (NYHA III, IV) (at any time), serious uncontrolled cardiac arrhythmia (at any time), myocardial infarction or cerebrovascular accidents ≤ 6 months prior to first study treatment or history of left ventricular dysfunction
* reduced left ventricular ejection fraction (LVEF) of <50% on screening with echocardiogram or multiple gates acquisition (MUGA) scan
* severe valvulopathies with documented compromise in cardiac function
* Any of the following on screening ECG:
* QTc interval > 480 msec (or family history of congenital QTc prolongation)
* Right bundle branch block + left anterior hemiblock (bifascicular block)
* Complete left bundle branch block
* Any conduction abnormality requiring pacemaker
* Symptomatic sinus bradycardia
* Any ventricular arrhythmia except for benign premature ventricular contractions
* Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
* Symptomatic pericarditis
* Documented cardiomyopathy of any cause
* Female patients who are pregnant or breast feeding; pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum βhCG laboratory test (> 5 mIU/mL).
* Patients unwilling or unable to comply with adequate double barrier contraception throughout the trial and for 12 weeks after the last dose of study drug (by both male and female patients). This includes the following considerations:
* Hormonal contraceptives may be affected by cytochrome P450 interactions, and are therefore considered neither indicated nor effective.
* Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper), sponge or spermicide.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL [for US only: and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Patients who have a history of another primary malignancy and are off treatment for ≤ 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of the uterine cervix.
* Patients who have received attenuated live vaccines within one week of study entry. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Known intolerance to the study drug (or any of the excipients), and/or known hypersensitivity to PI3K inhibitor (eg. GDC-0980), and/or known hypersensitivity to rapamycins (eg. Sirolimus, everolimus, temsirolimus) or any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Molina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Carlo MI, Molina AM, Lakhman Y, Patil S, Woo K, DeLuca J, Lee CH, Hsieh JJ, Feldman DR, Motzer RJ, Voss MH. A Phase Ib Study of BEZ235, a Dual Inhibitor of Phosphatidylinositol 3-Kinase (PI3K) and Mammalian Target of Rapamycin (mTOR), in Patients With Advanced Renal Cell Carcinoma. Oncologist. 2016 Jul;21(7):787-8. doi: 10.1634/theoncologist.2016-0145. Epub 2016 Jun 10. PMID 27286790
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: BEZ235 400mg: Cohort 1: BEZ235 400mg by mouth twice daily
- Cohort -1: BEZ235 200mg: Cohort -1: BEZ235 200mg by mouth twice daily
- Cohort -1a: BEZ235 300mg: Cohort -1a: BEZ235 300mg by mouth twice daily
Period: Overall Study
Arm/Group | Cohort 1: BEZ235 400mg | Cohort -1: BEZ235 200mg | Cohort -1a: BEZ235 300mg
Started | 2 | 6 | 2
Completed | 0 | 5 | 0
Not Completed | 2 | 1 | 2
Not completed — Dose Limiting Toxicity (DLT) | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: BEZ235 400mg | Cohort -1: BEZ235 200mg | Cohort -1a: BEZ235 300mg | Total
Number analyzed (Participants) | 2 | 6 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 1 | 6
  >=65 years | 2 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3
  Male | 2 | 4 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 2 | 6 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: In patients with advanced clear cell RCC, progressing after prior first-line or second-line mTOR therapy. The determination of antitumor efficacy will be based on objective tumor assessments made according to the RECIST1.1.
Time Frame: 1 year
Population: ORR was only assessed for participants who completed the study, which were only 5 patients on Cohort -1
Measure: Number; unit: participants
Arm/Group | Cohort -1: BEZ235 200mg
Number analyzed (Participants) | 5
participants
  Progression of Disease | 3
  Stable Disease | 2

ADVERSE EVENTS:
Arm/Group | Cohort 1: BEZ235 400mg | Cohort -1: BEZ235 200mg | Cohort -1a: BEZ235 300mg
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/6 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 3/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: BEZ235 400mg (N=2) | Cohort -1: BEZ235 200mg (N=6) | Cohort -1a: BEZ235 300mg (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: BEZ235 400mg (N=2) | Cohort -1: BEZ235 200mg (N=6) | Cohort -1a: BEZ235 300mg (N=2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Given the number of toxicities seen and the difficulty with patient retention in the dose escalation portion, the sponsor decided to close the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes